CLINICAL TRIAL: NCT04483765
Title: Does Shock Index, Modified Shock Index and Age-Related Shock Index Have a Predictive Value in Predicting the Risk of Post-spinal Hypotension in Elderly Patients
Brief Title: Shock Index, Modified Shock Index and Age-related Shock Index for Predicting Post-spinal Hypotension in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-20-787
Record Dates: First submitted 2020-07-18; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Anesthesia Morbidity; Procedural Hypotension; Intraoperative Hypotension; Geriatrics
Keywords: geriatric anesthesia; post-spinal hypotension; Intraoperative Hypotension; spinal anesthesia; shock index; modified shock index; age-related shock index
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post-spinal hypotension: Patients with a fall in SBP by 25% of the preoperative baseline or an absolute value <90 mm of Hg; MAP ≤65 mmHg after spinal anesthesia
  Interventions: Procedure: spinal anesthesia
- post-spinal normotension: Patients with Fall of SBP<%25 of the preoperative value or absolute value >90 mm Hg, MAP>65 mmHg
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — patients undergoing transurethral resection of the prostate (TURP) and transurethral resection of the bladder (TURB) surgery under spinal anesthesia.

SUMMARY:
Aim of this prospective observational study is to investigate whether shock index(SI), modified shock index(MSI) and age related shock index(ASI) have any predictive value in predicting post-spinal hypotension which may develop in patients over 65 years of age, who are planned to undergo transurethral resection of the prostate (TURP) and transurethral resection of the bladder (TURB) surgery under spinal anesthesia.

DETAILED DESCRIPTION:
During the aging process, many important changes occur in the cardiovascular system. In elderly patients undergoing surgery, systemic vascular resistance is generally high but accompanying dehydration is a very common condition. The hemodynamic status of these patients may be compromised during spinal anesthesia due to the decrease in both systemic vascular resistance (SVR) and cardiac preload. Intraoperative hypotension may develop after spinal anesthesia. Intraoperative hypotension can prolong hospital stay by causing serious complications, and it can significantly affect mortality rates. Predicting hypotension which may develop after spinal anesthesia, can save time to decide, prepare and apply preventive interventions.

Shock index (SI) has been defined as the ratio of heart rate (HR) to systolic blood pressure (SBP). SI is an easy and non-invasive marker used in hypovolemia and early diagnosis of shock. SI is usually <0.7. In case of acute hypovolemia and circulatory failure, this ratio increases. It has been stated that in critical patients, diastolic blood pressure (DBP) will drop earlier than SBP, and the mean blood pressure will be a more accurate marker to assess the severity of the disease. For this reason, the modified shock index (MSI), which is obtained by dividing the heart rate by the mean arterial pressure (MAP), has been defined. MSI> 1.3 indicates a hypodynamic state.

The Age Shock Index (ASI) is defined by multiplying SI by age. In trauma patients, this index has been shown to correlate with a higher mortality rate with an increase greater than 50. Since age affects the physiological reserve negatively, it has been stated that ASI is a better predictor of 48-hour mortality compared to heart rate, SBP or SI. In studies evaluating ASI, SI and MSI to predict post-intubation hypotension; pre-intubation SI, MSI, ASI values have been shown to be the independent predictors of post-intubation hypotension.

Aim of this prospective observational study is to investigate whether SI, MSI and ASI have any predictive value in predicting post-spinal hypotension which may develop in patients over 65 years of age, who are planned to undergo transurethral resection of the prostate (TURP) and transurethral resection of the bladder (TURB) surgery under spinal anesthesia.

The secondary objective is to compare the two groups in terms of preoperative and postoperative blood tests, and to determine whether the patients were admitted to intensive care or postanesthesia care unit. If the patient was admitted, length of unit and hospital stay and postoperative complications (if developed any) will be recorded. In addition, the investigators will examine whether intraoperative hypotension has any negative effects.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years old

Exclusion Criteria:

duration of operation>120 minutes ASA>3

* Patients with valvular heart disease that disrupts hemodynamics
* Patients with arrhythmia (such as atrial fibrillation with rapid ventricular rate) that disrupts hemodynamics
* severe heart failure
* mental and motor problems
* neuropsychiatric disorders

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Paients undergo transurethral resection of the prostate (TURP) and transurethral resection of the bladder (TURB) surgery under spinal anesthesia.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
SI | preoperative
  shock index: defined as the ratio of heart rate (HR) to systolic blood pressure (SBP)
MSI | preoperative
  Modified Shock İndex: obtained by dividing the heart rate by the mean arterial pressure
ASI | preoperative
  Age Shock Index (ASI) is defined by multiplying shock index(SI) by age

SECONDARY OUTCOMES:
CCI | preoperative
  Charlson Comorbidity Index
length of hospital stay | through study completion, an average of 3 months
  length of hospital stay after operation

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Aytac, Principal Investigator — Ankara City Hospital Anesthesiology Department
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No